CLINICAL TRIAL: NCT06943612
Title: Colorectal Resections and Reconstructions in Patients With Retroperitoneal Sarcoma: Evaluation of Surgical Strategies and Postoperative Quality of Life
Brief Title: Colorectal Resections in Patients With Retroperitoneal Sarcoma
Acronym: COLOSARC-Q
Status: Recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Jens Jakob, Head Sarcoma Surgery and Sarcoma Center Mannheim, Heidelberg University, Heidelberg University
Other Study IDs: 2024-562; DRKS00034135 (Other: German Register of Clinical Studies (DRKS))
Record Dates: First submitted 2025-04-10; First posted 2025-04-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma, Soft Tissue; Retroperitoneal Sarcoma
Keywords: Soft tissue sarcoma; Retroperitoneal Sarcoma; Sarcoma Surgery; Stoma; Colorectal resection
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary, retroperitoneal sarcomas who underwent surgery with colorectal resection: Patients with primary retroperitoneal sarcomas who underwent surgery with colorectal resection at DKG-certified sarcoma centers or hospitals in Germany and Switzerland that meet certification-equivalent criteria

SUMMARY:
COLOSARC-Q is a multicenter study with the objective of providing an up-to-date assessment of colorectal resections and reconstruction techniques in the context of multivisceral resections for retroperitoneal sarcomas, as well as colorectal surgery-associated complications and their impact on patients' quality of life.

In multivisceral resections involving the colon and rectum, the primary aim is to achieve complete resection and preserve organ function. However, multivisceral resections have a high risk of perioperative morbidity including anastomotic leakage. The proposed project aims to determine the number of primary anastomoses, their insufficiency rates, and the fraction of patients with primary and secondary stomas. In addition, the patients' quality of life after multivisceral sarcoma resection is to be recorded using standardized surveys.

The analysis has the potential to facilitate intraoperative decision-making for colorectal resections in the context of multivisceral resections.

DETAILED DESCRIPTION:
The primary goal of retroperitoneal sarcoma surgery is to achieve complete resection. The resection of retroperitoneal sarcomas (RPS) usually involves the removal of parts of the colon. While there is good data on surgical principles and postoperative complications of multivisceral resections in RPS as a whole (1, 2), there is little evidence on the frequency of temporary or permanent stomas and complications associated with intestinal surgery (e.g., number of anastomotic leackages in relation to the number of intestinal anastomoses performed) and their impact on the quality of life of those affected.

The COLOSARC-Q study is a multicenter, non-interventional study with the aim of documenting

* colorectal resection and reconstruction techniques in connection with multivisceral resections in retroperitoneal sarcomas (RPS),
* complications associated with intestinal surgery in multivisceral resections, and
* the resulting effects on the quality of life of sarcoma patients. The project plans to include 120 patients with retroperitoneal sarcomas who have undergone colon resection as part of a multivisceral resection at a DKG-certified sarcoma center or hospital that meets certification-equivalent criteria. For these patients, patient-, tumor-, and treatment-specific parameters (all patients), standardized questionnaires on health-related quality of life (EORTC QLQ - C30 (version 3.0)) and bowel function (EORTC QLQ - CR29) (expected response rate ≥ 50%) and semi-structured interviews with the aim of recording specific problems that may not be covered in the questionnaires (e.g., regarding stoma placement, nutritional status, treatment sequence, or home care; n = 10-15).

COLOSARC-Q has the potential to improve preoperative participatory decision-making and intraoperative strategy in colorectal resections as part of multivisceral resections in order to reduce complication rates and develop surgical strategies tailored to specific patient needs.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation with evidence of a retroperitoneal sarcoma
* Tumor resection with colorectal resection
* Surgery in a DKG-certified sarcoma center or hospital that meets certification-equivalent criteria
* Age 18 years or older
* Written consent

Exclusion Criteria:

* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary, retroperitoneal sarcomas who underwent surgery with colorectal resection at DKG-certified sarcoma centers or hospitals in Germany and Switzerland that meet certification-equivalent criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of resection and reconstruction procedures of the colon and rectum in the context of multivisceral resections of retroperitoneal sarcomas | immediately after the surgery
  Description of the surgical procedure, e.g. righ hemicolectomy with primary anastomosis

SECONDARY OUTCOMES:
Postoperative complications associated with resections and reconstructions of the bowel | up to 90 days after surgery
  Evaluation of postoperative complications associated with resections and reconstructions of the bowel during and after multivisceral resections of retroperitoneal sarcomas (Comprehensive Complication Index (CCI), up to 90 days postoperatively)
Assessment of quality of life after colorectal resections in the context of RPS resections | through study completion, an average of 1 year
  Assessment of quality of life after using the EORTC QLQ - C30 (Version 3.0) questionnaires)
Assessment of changes in bowel function after resection of retroperitoneal sarcomas | through study completion, an average of 1 year
  Assessment of the bowel function using the EORTC QLQ - CR29 questionnaire
Identification of problems and needs of RPS patients | through study completion, an average of 1 year
  Identification of problems and needs of RPS patients who have undergone resection and reconstruction of the colon, e.g. with regard to education, home care, bowel function, stoma care, rehabilitation measures and therapy intensity and sequence
Determination of patient-, tumor- and treatment-related factors influencing the above-mentioned primary and secondary study objectives | through study completion, an average of 1 year
  Determination of the influence of the following patient-, tumor- and treatment-related factors on the above-mentioned primary and secondary study objectives:
  * Gender
  * age
  * Body mass index (BMI)
  * Malnutrition (serum albumin preoperatively)
  * Concomitant diseases (e.g. diabetes mellitus, coronary heart disease)
  * Previous abdominal surgery
  * Size, localization (left/right), grading and histological subtype of the RPS
  * Neoadjuvant therapies (radiotherapy and/or chemotherapy)
  * Operation time
  * Intraoperative blood loss
  * Extent of the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jens Jakob, Prof., Principal Investigator — Sarcoma Unit, Department of Surgery, University Medical Center Mannheim, Theodor-Kutzer-Ufer 1-3, 68167 Mannheim, Germany
Locations (13):
- Germany (12):
  - Sarcoma Center of University Medical Center Mannheim, Mannheim, Baden-Wurttemberg
  - Helios Hospital Berlin-Buch, Berlin
  - University Medical Center Dresden, Dresden
  - University Medical Center Erlangen, Erlangen
  - University Medical Center Halle, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medical University of Hannover, Hanover
  - Heidelberg University Hospital, Heidelberg
  - University Hospital Magdeburg, Magdeburg
  - LMU Hospital, München
  - University Medical Center Tübingen, Tübingen
  - University Medical Center Ulm, Ulm
- Sarcoma Center University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakob J, Hentschel L, Richter S, Kreisel I, Hohenberger P, Kasper B, Andreou D, Pink D, Schmitt J, Schuler MK, Eichler M. Transferability of Health-Related Quality of Life Data of Large Observational Studies to Clinical Practice: Comparing Retroperitoneal Sarcoma Patients from the PROSa Study to a TARPS-WG Cohort. Oncol Res Treat. 2022;45(11):660-669. doi: 10.1159/000525288. Epub 2022 Jun 14. PMID 35700716
- [Background] MacNeill AJ, Fiore M. Surgical morbidity in retroperitoneal sarcoma resection. J Surg Oncol. 2018 Jan;117(1):56-61. doi: 10.1002/jso.24902. Epub 2018 Jan 3. PMID 29314041
- [Background] Bonvalot S, Raut CP, Pollock RE, Rutkowski P, Strauss DC, Hayes AJ, Van Coevorden F, Fiore M, Stoeckle E, Hohenberger P, Gronchi A. Technical considerations in surgery for retroperitoneal sarcomas: position paper from E-Surge, a master class in sarcoma surgery, and EORTC-STBSG. Ann Surg Oncol. 2012 Sep;19(9):2981-91. doi: 10.1245/s10434-012-2342-2. Epub 2012 Apr 3. PMID 22476756
- [Background] Gronchi A, Strauss DC, Miceli R, Bonvalot S, Swallow CJ, Hohenberger P, Van Coevorden F, Rutkowski P, Callegaro D, Hayes AJ, Honore C, Fairweather M, Cannell A, Jakob J, Haas RL, Szacht M, Fiore M, Casali PG, Pollock RE, Raut CP. Variability in Patterns of Recurrence After Resection of Primary Retroperitoneal Sarcoma (RPS): A Report on 1007 Patients From the Multi-institutional Collaborative RPS Working Group. Ann Surg. 2016 May;263(5):1002-9. doi: 10.1097/SLA.0000000000001447. PMID 26727100
- [Derived] Hettler M, Scharpf KR, Eich A, Albertsmeier M, Dupree A, Hetjens S, Harbrucker M, Menge F, Betzler A, Hohenberger P, Jakob J. Multicentre prospective non-interventional study protocol for evaluating surgical strategies for Colorectal Resections and Postoperative Quality of Life in Retroperitoneal Sarcoma Patients Across German-Speaking Sarcoma Centres (COLOSARC-Q). BMJ Open. 2025 Dec 30;15(12):e102015. doi: 10.1136/bmjopen-2025-102015. PMID 41469069
- See also: The study is supported by the Association of Surgical Oncology of the German Surgical Society that provides some information on the study on their website — https://www.aco-chirurgie.de/kollegen/forschung/